CLINICAL TRIAL: NCT00504686
Title: Validation of a Clinical Prediction Rule to Identify Patients With Neck Pain Likely to Benefit From Thoracic Spine Thrust Mobilization: A Randomized Clinical Trial
Brief Title: Patients With Neck Pain Likely to Benefit From Thoracic Spine Thrust Mobilization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Collaborators: Newton-Wellesley Hospital (Other)
Responsible Party: Joshua Cleland, Franklin Pierce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC 06-14
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): manual therapy - thoracic spine thrust manipulation
  Interventions: Other: manual therapy; Other: exercise
- 2 (Active Comparator): therapeutic exercise
  Interventions: Other: exercise

INTERVENTIONS:
Other: manual therapy — manual therapy - thoracic spine thrust manipulation
  Arms: 1
Other: exercise — therapeutic exercise

SUMMARY:
Recently a clinical prediction rule (CPR) has been developed that identifies patients with neck pain who are likely to respond rapidly and dramatically to thoracic spine thrust manipulation and an active range of motion exercise. Although the initial predictor variables identified during the development of a thoracic spine manipulation CPR seem to have adequate face validity, there is no guarantee that these factors will persist in a different group of patients, even ones with similar characteristics as those used in the initial exploratory study. The purpose of this follow-up study in which patients will be randomly assigned to receive thoracic spine thrust manipulation followed by therapeutic exercises or therapeutic exercise alone will be to investigate the validity of the previously developed CPR. If the CPR is indeed meaningful, patients who are positive on the CPR and receive thoracic spine thrust manipulation should experience improved outcomes compared to patients who are negative on the CPR and receive thoracic spine manipulation, and compared to patients who are positive on the CPR but receive the intervention believed to be effective for another subgroup of patients with neck pain.

DETAILED DESCRIPTION:
Background: Recently a clinical prediction rule (CPR) has been developed that identifies patients with neck pain who are likely to respond rapidly and dramatically to thoracic spine thrust manipulation and an active range of motion exercise. Although the initial predictor variables identified during the development of a thoracic spine manipulation CPR seem to have adequate face validity, there is no guarantee that these factors will persist in a different group of patients, even ones with similar characteristics as those used in the initial exploratory study.

Purpose: The purpose of this follow-up study in which patients will be randomly assigned to receive thoracic spine thrust manipulation followed by therapeutic exercises or therapeutic exercise alone will be to investigate the validity of the previously developed CPR. If the CPR is indeed meaningful, patients who are positive on the CPR and receive thoracic spine thrust manipulation should experience improved outcomes compared to patients who are negative on the CPR and receive thoracic spine manipulation, and compared to patients who are positive on the CPR but receive the intervention believed to be effective for another subgroup of patients with neck pain.

Design: We will conduct a multi-center randomized clinical trial to assess the effectiveness of a previously-developed CPR for identifying patients with neck pain likely to respond to a thoracic spine thrust manipulation. Subjects between the ages of 18 and 60 with a primary report of neck pain will be randomized to receive manipulation plus an exercise program or to receive an exercise program only.

Methods: One hundred and forty patients with a primary complaint of neck pain who meet the inclusion/exclusion criteria and consent to participate will be enrolled in the study. We based sample size calculations on detecting a statistically significant difference between any of the 4 cells of the study which include the patients status on the rule (patients that meet the CPR and patients that do not meet the CPR) and treatment group (manipulation and exercise) by using the 1-week Neck Disability Index (NDI) score at an alpha-level of 0.05. To detect a 10 point change in NDI, with an expected standard deviation of 12 points at the 1 week follow up (effect size 0.80) with 90% power using a two-tailed hypothesis and assuming a 50% distribution of patients who do and do not meet the rule, 31 patients per cell are required. We will recruit 140 subjects into the study to control for drop-outs prior to the 1 and 4 week follow-up and possible distribution discrepancies between the classifications. The primary outcome point is four-weeks after randomization, with change in disability as measured by the NDI, serving as the primary outcome measure.

Data Analysis: We will examine the primary aim with a 3-way repeated-measures analysis of variance (ANOVA) with treatment group (manipulation vs. exercise) and status on the rule (positive or negative) as the between subjects independent variables and time (baseline, 1 week and 4 weeks) as the within-subjects independent variable. The dependent variable will be disability (NDI score). The hypothesis of interest is the 3-way group * CPR status * time interaction. We will perform planned pairwise comparisons at each follow-up period by using the Bonferroni inequality.

Significance: The results of this study should improve clinical decision-making and outcomes from physical therapy intervention by assisting clinicians in their ability to select appropriate manual physical therapy techniques for patients with neck pain. Validation of the CPR would enhance the certainty in which therapists will be able to identify patients with neck pain who are likely to exhibit a dramatic response to thoracic spine thrust manipulation as measured by reduced levels of disability) and therapeutic exercises. Results of the study will impact future patients with neck pain as it will provide a method of classification in which based on their clinical presentation therapists can determine the likelihood that they will or will not respond to thoracic spine thrust manipulation.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria will be used to determine eligibility for this study:

1. Primary complaint of neck pain with or without unilateral upper extremity symptoms
2. Age between 18-60 years old
3. NDI score greater than 10 points

Exclusion Criteria:

The following exclusion criteria will be used to determine ineligibility for this study:

1. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
2. History of whiplash injury within the past six weeks
3. Diagnosis of cervical spinal stenosis or bilateral upper extremity symptoms
4. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:
6. Muscle weakness involving a major muscle group of the upper extremity
7. Diminished upper extremity muscle stretch reflex (biceps brachii, brachioradialis, or triceps reflex)
8. Diminished or absent sensation to pinprick in any upper extremity dermatome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 4 weeks, 6 months

SECONDARY OUTCOMES:
Pain | 4 week, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joshua A Cleland, PT, PhD, Principal Investigator — Franklin Pierce University
Locations (1):
- Concord Hospital, Concord, New Hampshire, United States

REFERENCES:
- [Derived] Cleland JA, Mintken PE, Carpenter K, Fritz JM, Glynn P, Whitman J, Childs JD. Examination of a clinical prediction rule to identify patients with neck pain likely to benefit from thoracic spine thrust manipulation and a general cervical range of motion exercise: multi-center randomized clinical trial. Phys Ther. 2010 Sep;90(9):1239-50. doi: 10.2522/ptj.20100123. Epub 2010 Jul 15. PMID 20634268